CLINICAL TRIAL: NCT06309966
Title: A Phase 2/3 Multicenter, Randomization, Double-Blind, Placebo-Controlled, Study to Evaluate the Efficacy, Safety and Tolerability of BHV-7000 in Subjects With Refractory Focal Onset Epilepsy
Brief Title: Study to Determine if BHV-7000 is Effective and Safe in Adults With Refractory Focal Onset Epilepsy
Acronym: RISE 3
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV7000-303; 2023-508811-21 (Registry Identifier: EU CTR)
Record Dates: First submitted 2024-03-08; First posted 2024-03-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Focal Epilepsy
Keywords: Focal Epilepsy; Epilepsy; Seizure; Refractory Epilepsy; Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures; Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BHV-7000 50 mg (Experimental)
  Interventions: Drug: BHV-7000
- BHV-7000 75 mg (Experimental)
  Interventions: Drug: BHV-7000
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 50 mg. Participants will take blinded investigational product (IP) once daily
  Arms: BHV-7000 50 mg
Drug: BHV-7000 — BHV-7000 75 mg. Participants will take blinded investigational product (IP) once daily
  Arms: BHV-7000 75 mg
Drug: Placebo — Matching placebo taken once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether BHV-7000 is effective in the treatment of refractory focal epilepsy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and Female participants 18 to 75 years of age at time of consent.
2. Diagnosis of Focal Onset Epilepsy at least 1 year prior to screening visit defined by 2017 International League Against Epilepsy (ILAE) Classification and based on requirements of Epilepsy Adjudication criteria.

   a. Focal seizures i. Focal aware seizures with clinically observable signs and/or symptoms ii. Focal impaired awareness seizures with clinically observable signs and/or symptoms iii. Focal to bilateral tonic-clonic seizures
3. Subject meets the 2009 ILAE definition of drug resistant epilepsy, failure of adequate trials of two tolerated and appropriately chosen and used anti-seizure medication (ASM) schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom.
4. Ability to keep accurate seizure diaries
5. Current treatment with at least 1 and up to 3 ASMs and 4 epilepsy treatments in total

Key Exclusion Criteria:

1. History of status epilepticus (convulsive status epilepticus for > 5 minutes or focal status epilepticus with impaired consciousness for > 10 minutes) within the last 6 months prior to screening visit that is not consistent with the subject's habitual seizure.
2. History of repetitive/cluster seizures (where individual seizures cannot be counted) within the last 6 months prior to screening visit and during observation phase.
3. Resection neurosurgery for seizures <4 months prior to the screening visit.
4. Radiosurgery performed <2 years prior to the screening visit.
5. Subjects with only focal aware nonmotor seizures which involve subjective sensory or psychic phenomena only, without impairment of consciousness or awareness (formally called simple partial seizures), with or without ictal EEG correlation with clinical symptoms.
6. Any condition that would interfere with the subject's ability to comply with study instructions, place the subject at unacceptable risk, and/or confound the interpretation of safety or efficacy data from the study, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 28-day average seizure frequency | Baseline, Week 8 to Week 16
  To compare the efficacy of each of 2 doses of BHV-7000 to placebo as an adjunctive therapy for refractory focal onset epilepsy as measured by the change from OP (observational phase) in 28-day average seizure frequency. The primary objective will be measured by comparing the observation phase (8 weeks) to the 8-week double-blind treatment phase.

SECONDARY OUTCOMES:
Percentage of Participants with at at least 50% reduction in seizure frequency per month | Baseline, Week 8 to Week 16
  To compare the efficacy of 2 dose strengths of BHV-7000 to placebo as adjunctive therapy for refractory focal onset epilepsy as measured by the proportion of subjects that have at least a 50% reduction in seizures per month (28 days). This objective will be measured by comparing the proportion of subjects with at least a 50% reduction in 28-day average seizure frequency over the course of the 8 week double-blind phase to the observation phase.
Change from Baseline in 28-day average seizure frequency during first month of treatment | Baseline, Week 8 to Week 12
  To compare the efficacy of BHV-7000 to placebo during the first month of treatment. This objective will be measured by the change in log-transformed 28-day adjusted seizure frequency from observation phase over the first month of the double blind phase.
Percentage of Participants with at at least 75% reduction in seizure frequency per month | Baseline, Week 8 to Week 16
  To compare the efficacy of BHV-7000 to placebo as measured by the proportion of subjects that have at least a 75% reduction in seizures per month (28 days). This objective will be measured by comparing the proportion of subjects with at least a 75% reduction in 28-day average seizure frequency over the course of the double-blind phase compared to the observation phase.
Percentage of Participants with seizure freedom during DB Phase | Week 8 to Week 16
  To compare the efficacy of BHV-7000 to placebo on seizure freedom (100% seizure reduction during the DBP phase). This objective will be measured by proportion of subjects that are seizure free during the double-blind phase.
Change from baseline in 7-day adjusted seizure frequency during first week of treatment | Baseline, Week 8 to Week 9
  To compare the efficacy of BHV-7000 to placebo during the first week of treatment. This objective will be measured by the change in log-transformed 7-day adjusted seziure frequency from observation phase over the first week of the double-blind phase.
Change from baseline in Patient Global Impression of Change (PGI-C) | Baseline, Week 16
  To compare the efficacy of BHV-7000 to placebo on the patient global impression of change (PGI-C). This objective will be measured by proportion of subjects at week 8 of double-blind treatment phase with a PGI-C response of "minimally improved", "much improved" or "very much improved". This scale is a 7-point Likert scale with response options of:
  (1) "very much improved" , (2) "much improved", (3) "minimally improved", (4) "no change", (5) "minimally worse", (6) "much worse", (7) and "very much worse"
Number of Participants With Deaths, Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and moderate or severe AEs | Week 8 to Week 16
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with deaths, SAEs, AEs leading to discontinuation, and moderate and severe AEs.
Number of Participants With Clinically Significant Laboratory Abnormalities | Week 8 to Week 16
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 or 4 laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (172):
- United States (66):
  - Accel Research, Birmingham, Alabama
  - Onyx Clinical Trials, Peoria, Arizona
  - Xenoscience, Inc., Phoenix, Arizona
  - University of Arizona / Banner University Medical Center Phoenix, Phoenix, Arizona
  - ARENSIA Exploratory Medicine, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Amicis Research Center, Lancaster, California
  - Memorialcare Miller Children's & Women's Hospital Long Beach, Long Beach, California
  - Tri Valley Neurology Medical Associates, Inc., Mission Hills, California
  - Stanford University, Palo Alto, California
  - Profound Research LLC, Poway, California
  - Kaiser Permanente, Aurora, Colorado
  - UConn Health, Farmington, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - EZR Research, LLC, Boca Raton, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Las Mercedes Medical Research, Hialeah, Florida
  - Coral Clinic Research, Homestead, Florida
  - Dm Healthworks, Kissimmee, Florida
  - Y&L Advance Health Care, Inc d/b/a Elite Clinical Research, Miami, Florida
  - Serenity Research Center, Miami, Florida
  - Research Institute of Orlando, Orlando, Florida
  - Comprehensive Neurology Clinic, Orlando, Florida
  - Panhandle Research & Medical Clinic, Pensacola, Florida
  - Knight Neurology, Rockledge, Florida
  - PENS, Tampa, Florida
  - Encore Medical Research of Weston LLC., Weston, Florida
  - Accelerated Clinical Trials, LLC, Peachtree Corners, Georgia
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - OLORMC, Baton Rouge, Louisiana
  - DelRicht Research, Baton Rouge, Louisiana
  - Neurocare Of Louisiana, Covington, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - LSU Health Shreveport, Shreveport, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Boston Neuro Research, South Dartmouth, Massachusetts
  - SRI International, Plymouth, Michigan
  - University of Missouri Health Care, Columbia, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - NEREG, Hackensack, New Jersey
  - Tekton Research, Marlboro, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - Northwell Health, Great Neck, New York
  - Northwell Health Ped. Neurology, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - Cincinatti Children's Hospital, Cincinnati, Ohio
  - Wright State University, Dayton, Ohio
  - Oregon Neurology Associates, Springfield, Oregon
  - AHN, Pittsburgh, Pennsylvania
  - MUSC, Charleston, South Carolina
  - WR-ClinSearch, Chattanooga, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Horizon Clinical Research Group, Cypress, Texas
  - M3 Wake Research-Dallas, Dallas, Texas
  - ANESC Research, El Paso, Texas
  - Tarrant Neurology Associates, Fort Worth, Texas
  - UTHealth Houston, Houston, Texas
  - UTHSC, Houston, Texas
  - Stryde Research, Plano, Texas
  - Intermountain Health, Murray, Utah
  - Medstar Health Research Institute, McLean, Virginia
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - St Vincents Hospital Melbourne - PPDS, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Flinders Medical Centre, Bedford Park
- Denmark (3):
  - Odense Universitetshospital, Odense, Fyn
  - Aarhus University Hospital, Aarhus
  - Epilepsihospitalet Filadelfia, Dianalund
- Finland (3):
  - Kuopion yliopistollinen sairaala, Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Helsinki University Hospital, Helsinki, Uusimaa
- Germany (16):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Epilepsiezentrum Kork, Kehl, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - LMU Klinikum der Universität München - Campus Großhadern, München, Bavaria
  - Epilepsieklinik Tabor, Bernau bei Berlin, Brandenburg
  - Universitätsklinikum Gießen und Marburg GmbH - Standort Marburg, Marburg, Hesse
  - Klinikum Osnabrück GmbH, Osnabrück, Lower Saxony
  - Krankenhaus Mara gGmbH, Bielefeld, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Kleinwachau Sächsisches Epilepsiezentrum Radeberg Gemeinnützige Gmbh, Radeberg, Saxony
  - Vivantes - Humboldt Klinikum, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Epilepsie-Zentrum Bodensee, Ravensburg
- Greece (5):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - University General Hospital ''ATTIKON'', Chaïdári
  - University General Hospital of Ioannina, Ioannina
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Semmel Egyet Idegsebésze Neuro Klin, Budapest, Hungary
- India (5):
  - Nizam's Insti. of Medical Sciences, Hyderabad
  - Mallikatta Neuro Centre, Mangalore
  - Jaslok Hospital and Research, Mumbai
  - Dr G M Taori Memorial CIIMS, Nagpur
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Italy (17):
  - Università degli Studi G. D'Annunzio Chieti-Pescara, Chieti, Abruzzo
  - Azienda Ospedaliera Universitaria Renato Dulbecco - AO Mater Domini, Catanzaro, Calabria
  - AORN Antonio Cardarelli, Napoli, Campania
  - AUSL di Bologna - Ospedale Bellaria, Bologna, Emilia-Romagna
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genoa, Liguria
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - ASST Santi Paolo e Carlo - Azienda Universitaria-Polo Universitario San Paolo, Milan, Lombardy
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero-Universitaria di Modena - Ospedale Civile di Baggiovara, Baggiovara, Modena
  - IRCCS Istituto Neurologico Mediterraneo Neuromed, Pozzilli, Molise
  - Università Politecnica delle Marche Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona, The Marches
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Calambrone, Tuscany
  - Fondazione Policlinico Universitario A Gemelli-Rome, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Rome
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona
- Mexico (7):
  - Unidad de Investigación en Salud de Chihuahua S.C.-Mexico city, Mexico City
  - Clinstile, S.A. de C.V., Mexico City
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey
  - Axis Heilsa S. de R.L. de C.V., Obispado
  - Neurociencias Estudios Clinicos S.C., Sinaloa
  - Clinical Research Institute SC-Mexico, Tlalnepantla
  - FAICIC S De RL De CV, Veracruz
- Poland (5):
  - MTZ Clinical Research, Krakow
  - Pratia MCM Krakow, Krakow
  - LANDA Specjalistyczne, Krakow
  - Neurosphera SP. Z O.O, Warsaw
  - Premium Clinic Wrocław, Wroclaw
- Portugal (6):
  - ULS de Entre Douro e Vouga, EPE - Hospital de São Sebastião, Santa Maria da Feira, Aveiro District
  - ULS de Matosinhos, EPE - Hospital Pedro Hispano, Senhora da Hora, Porto District
  - Centro Clínico Académico, Braga - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Hospital da Luz Torres de Lisboa, Lisbon
- Romania (2):
  - Targu-Mures Emergency Clinical County Hospital - Str. Gh. Marinescu nr.50, Târgu Mureş, Mureș County
  - Emergency University Hospital, Bucharest
- Slovakia (2):
  - IN MEDIC, s.r.o., Bardejov
  - Kraskova 2636, Neurologické oddelenie, Rimavská Sobota
- Spain (18):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Fundacio Assistencial Mutua de Terrassa, Barcelona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Vithas Granada, Granada
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Ruber Internacional (Grupo Quironsalud), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Blua Sanitas Valdebebas Hospital, Madrid
  - Hospital blua sanitas valdebebas, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Centro de Neurologia Avanzada, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- United Kingdom (8):
  - Morriston Hospital, Swansea, Glamorgan
  - Queen Elizabeth University Hospital-PPDS, Glasgow, Glasgow City
  - Salford Royal Hospital - PPDS, Salford, Manchester
  - The Walton Centre - PPDS, Liverpool, Merseyside
  - University College London Hospitals (UCLH), London, Middlesex
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - University Hospital of Wales, Cardiff, South Glamorgan
  - Royal Victoria Infirmary, Newcastle upon Tyne